CLINICAL TRIAL: NCT03684642
Title: A 56-week, Multicenter, Open-label, Active-controlled, Randomized Study to Evaluate the Efficacy and Safety of Efpeglenatide Once Weekly Compared to Dulaglutide Once Weekly in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin
Brief Title: Efficacy and Safety of Efpeglenatide Versus Dulaglutide in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin
Acronym: AMPLITUDE-D
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to cancel TRIAL, not related to safety concern.
Sponsor: Sanofi (Industry)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC14829; 2017-002956-10 (EudraCT Number); U1111-1205-3150 (Other: UTN)
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — efpeglenatide; dulaglutide

STUDY DESIGN:
Masking Description: The study was open-label for the tested versus comparator drug and double blind for the doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efpeglenatide 4 mg (Experimental): Participants received Efpeglenatide subcutaneous (SC) injection once weekly up to Week 56 on top of metformin. Participants initiated dosing at 2 mg once weekly and increased every 2 weeks to the maximum of 4 mg once weekly for the treatment duration.
  Interventions: Drug: Efpeglenatide; Drug: Background therapy Metformin
- Efpeglenatide 6 mg (Experimental): Participants received Efpeglenatide SC injection once weekly up to Week 56 on top of metformin. Participants initiated dosing at 2 mg once weekly and increased every 2 weeks to the maximum of 6 mg once weekly for the treatment duration.
  Interventions: Drug: Efpeglenatide; Drug: Background therapy Metformin
- Dulaglutide 1.5 mg (Active Comparator): Participants received Dulaglutide SC injection once weekly up to Week 56 on top of metformin. Participants initiated dosing at 0.75 mg once weekly and increased after 2 weeks to 1.5 mg once weekly for the treatment duration.
  Interventions: Drug: Dulaglutide; Drug: Background therapy Metformin

INTERVENTIONS:
Drug: Efpeglenatide — Pharmaceutical form: solution for injection; Route of administration: SC
  Other Names: SAR439977
  Arms: Efpeglenatide 4 mg; Efpeglenatide 6 mg
Drug: Dulaglutide — Pharmaceutical form: solution for injection; Route of administration: SC
  Other Names: Trulicity™
  Arms: Dulaglutide 1.5 mg
Drug: Background therapy Metformin — Pharmaceutical form: tablet; Route of administration: oral; Dose to be kept stable throughout the study.

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of once weekly injection of efpeglenatide in comparison to once weekly injection of dulaglutide on glycated hemoglobin (HbA1c) change in participants with Type 2 diabetes mellitus (T2DM) inadequately controlled with metformin.

Secondary Objectives:

* To demonstrate the superiority of once weekly injection of efpeglenatide with once weekly injection of dulaglutide on glycemic control.
* To demonstrate the superiority of once weekly injection of efpeglenatide with once weekly injection of dulaglutide on body weight.
* To evaluate the safety of once weekly injection of efpeglenatide and once weekly injection of dulaglutide.

DETAILED DESCRIPTION:
Study duration per participant was approximately 65 weeks including an up to 3-week Screening Period, a 56-week Treatment Period and a 6-week safety Follow-up Period.

ELIGIBILITY:
Inclusion criteria:

* Participant must be greater than or equal to (>=) 18 years of age at the time of signing the informed consent.
* Participants with T2DM.
* Diabetes diagnosed at least 1 year before screening.
* Participants on stable dose of at least 1500 milligram per day (mg/day) of metformin, or tolerated maximum dose, or as per country regulation if less, for at least 3 months prior to screening.
* HbA1c between 7.0 percent (%) and 10.0% (inclusive) measured by the central laboratory at screening.

Exclusion criteria:

* Retinopathy or maculopathy with one of the following treatments, either recent (within 3 months prior to screening) or planned: intravitreal injections or laser or vitrectomy surgery.
* Clinically relevant history of gastrointestinal (GI) disease associated with prolonged nausea and vomiting, including (but not limited to) gastroparesis, unstable and not controlled gastroesophageal reflux disease requiring medical treatment within 6 months prior to screening or history of surgery affecting gastric emptying.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy had been performed), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy.
* Personal or family history of medullary thyroid cancer (MTC) or genetic conditions that predisposes to MTC (e.g., multiple endocrine neoplasia syndromes).
* Body weight change of greater than or equal to (>=) 5 kilogram within the last 3 months prior to screening.
* Systolic blood pressure greater than (>)180 millimeter of mercury (mmHg) and/or diastolic blood pressure >100 mmHg at randomization.
* Severe renal disease as defined by estimated glomerular filtration rate (eGFR), by Modification of Diet in Renal Disease (MDRD)] of less than (<)30 mL/min/1.73 m^2.
* Laboratory findings at the screening visit:
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 * upper limit of normal (ULN) or total bilirubin >1.5 * ULN (except in case of documented Gilbert's syndrome);
* Amylase and/or lipase: >3 * ULN;
* Calcitonin >=5.9 picomoles per liter (pmol/L) (20 picograms per milliliter).
* Gastric surgery or other gastric procedures intended for weight loss within 2 years prior to screening, or planned during study period.
* Pregnant (confirmed by serum pregnancy test at screening) or breast-feeding women.
* Women of childbearing potential (WOCBP) not willing to use highly effective method(s) of birth control or who are unwilling to be tested for pregnancy during the study period and for at least 5 weeks after the last dose of study intervention.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (45):
- United States (30):
  - Investigational Site Number 8400038, Birmingham, Alabama
  - Investigational Site Number 8400035, Chandler, Arizona
  - Investigational Site Number 8400005, Glendale, Arizona
  - Investigational Site Number 8400054, Peoria, Arizona
  - Investigational Site Number 8400057, Huntington Park, California
  - Investigational Site Number 8400009, Los Angeles, California
  - Investigational Site Number 8400007, San Diego, California
  - Investigational Site Number 8400045, Spring Valley, California
  - Investigational Site Number 8400040, Tustin, California
  - Investigational Site Number 8400026, Van Nuys, California
  - Investigational Site Number 8400050, Waterbury, Connecticut
  - Investigational Site Number 8400055, Orlando, Florida
  - Investigational Site Number 8400041, Pembroke Pines, Florida
  - Investigational Site Number 8400025, Lawrenceville, Georgia
  - Investigational Site Number 8400060, Meridian, Idaho
  - Investigational Site Number 8400059, Skokie, Illinois
  - Investigational Site Number 8400044, Lexington, Kentucky
  - Investigational Site Number 8400061, Boston, Massachusetts
  - Investigational Site Number 8400001, Bridgeton, New Jersey
  - Investigational Site Number 8400039, New Windsor, New York
  - Investigational Site Number 8400028, Burlington, North Carolina
  - Investigational Site Number 8400036, Morehead City, North Carolina
  - Investigational Site Number 8400013, Maumee, Ohio
  - Investigational Site Number 8400014, Goose Creek, South Carolina
  - Investigational Site Number 8400030, Dallas, Texas
  - Investigational Site Number 8400020, San Antonio, Texas
  - Investigational Site Number 8400043, San Antonio, Texas
  - Investigational Site Number 8400053, San Antonio, Texas
  - Investigational Site Number 8400037, Layton, Utah
  - Investigational Site Number 8400049, Manassas, Virginia
- Hungary (5):
  - Investigational Site Number 3480004, Budapest
  - Investigational Site Number 3480003, Debrecen
  - Investigational Site Number 3480001, Gyula
  - Investigational Site Number 3480005, Hatvan
  - Investigational Site Number 3480002, Nyíregyháza
- Poland (6):
  - Investigational Site Number 6160008, Gdansk
  - Investigational Site Number 6160004, Gdynia
  - Investigational Site Number 6160010, Katowice
  - Investigational Site Number 6160009, Poznan
  - Investigational Site Number 6160003, Warsaw
  - Investigational Site Number 6160001, Wroclaw
- Ukraine (4):
  - Investigational Site Number 8040003, Kyiv
  - Investigational Site Number 8040001, Kyiv
  - Investigational Site Number 8040002, Kyiv
  - Investigational Site Number 8040004, Vinnytsia

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) by SANOFI: Product rights transferred to Hanmi Pharmaceutical.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 45 active sites in 4 countries. A total of 1608 participants were screened between 26 September 2018 and 17 December 2019, out of which 700 were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: A total of 908 participants were randomized in 1:1:1 ratio to either efpeglenatide 4 milligram (mg), efpeglenatide 6 mg, or dulaglutide 1.5 mg treatment arms, stratified by screening glycated hemoglobin (HbA1c) values (less than [<]8%, greater than or equal to [>=]8 percent [%]) and by body mass index (BMI) (<30 kg/m^2 and >=30 kg/m^2) on Day 1.
Period: Overall Study
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
Started | 303 | 302 | 303
Treated | 303 | 302 | 302
Safety Population (Participants who received at least 1 dose or part of a dose of the Investigational Medicinal Product (IMP), analyzed according to the treatment actually received.) | 313 (For safety analysis participants are included in the treatment group that they are exposed for longer duration. 10 participants randomized to Efpeglenatide 6 mg received 4 mg dose for longer duration, and considered in the Efpeglenatide 4 mg group for safety analysis.) | 292 | 302
Completed | 200 | 169 | 197
Not Completed | 103 | 133 | 106
Not completed — Adverse Event | 6 | 15 | 11
Not completed — Withdrawal by Subject | 35 | 53 | 23
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Poor compliance to protocol | 0 | 4 | 1
Not completed — Other than specified | 62 | 60 | 67
Not completed — Randomized and not treated | 0 | 0 | 1
Not completed — Missing completion status but alive at last contact | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat (ITT) population, which included all randomized participants, analyzed according to the treatment group allocated by randomization.
Groups:
- Efpeglenatide 4 mg: Participants received Efpeglenatide SC injection once weekly up to Week 56 on top of metformin. Participants initiated dosing at 2 mg once weekly and increased every 2 weeks to the maximum of 4 mg once weekly for the treatment duration.
- Total: Total of all reporting groups
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg | Total
Number analyzed (Participants) | 303 | 302 | 303 | 908
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.6) | 60.0 (10.1) | 59.4 (10.1) | 59.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 157 | 153 | 452
  Male | 161 | 145 | 150 | 456
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 271 | 263 | 275 | 809
  Black or African American | 24 | 30 | 18 | 72
  Asian | 5 | 3 | 6 | 14
  Other | 3 | 4 | 2 | 9
  Not reported | 0 | 2 | 2 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 33.4 (6.1) | 33.4 (6.2) | 33.4 (6.4) | 33.4 (6.2)
Baseline Glycated Hemoglobin (HbA1c %) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.12 (0.82) | 8.07 (0.78) | 8.11 (0.81) | 8.10 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 56 in HbA1c
Description: Adjusted Least square (LS) means and Standard errors (SE) were obtained from analysis of covariance (ANCOVA) model to account for missing data. Missing values were imputed by baseline observation carried forward (BOCF)-like multiple imputation method.
Time Frame: Baseline to Week 56
Population: Analysis was performed on modified intent-to-treat (mITT) population which included participants who completed study treatment; or who discontinued study treatment and completed/discontinued study before early termination; or who discontinued treatment before early termination and discontinued study due to early termination; or who discontinued treatment due to early termination within 30 days of target Week 56 visit.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 257 | 254 | 250
percentage of HbA1c | -1.12 (0.06) | -1.17 (0.06) | -1.09 (0.06)
Statistical Analysis 1: Comparison: Efpeglenatide 4 mg vs Dulaglutide 1.5 mg; A hierarchical step-down testing procedure was used to control type 1 error. Analysis was performed using ANCOVA model with the treatment groups, randomization strata, and geographical region as fixed classification effects, and baseline HbA1c value as a continuous covariate; Test type: Non-Inferiority — Non-inferiority of Efpeglenatide vs. Dulaglutide was demonstrated if the upper bound of the two-sided 95% confidence interval (CI) for the difference between groups was <=0.3%; Least Square (LS) Mean difference = -0.03, 95% CI 2-sided [-0.20 to 0.14], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Efpeglenatide 6 mg vs Dulaglutide 1.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority of Efpeglenatide vs. Dulaglutide was demonstrated if the upper bound of the two-sided 95% CI for the difference between groups was <=0.3%; LS Mean Difference = -0.08, 95% CI 2-sided [-0.25 to 0.09], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Efpeglenatide 4 mg vs Dulaglutide 1.5 mg; Test type: Superiority; p = 0.7064, ANCOVA — Threshold for significance at the level of 0.05
Statistical Analysis 4: Comparison: Efpeglenatide 6 mg vs Dulaglutide 1.5 mg; Test type: Superiority; p = 0.3427, ANCOVA — Threshold for significance at the level of 0.05

2. Secondary Outcome: Change From Baseline to Week 56 in Body Weight
Description: Adjusted LS means and SE were obtained from ANCOVA model to account for missing data. Missing values were imputed by BOCF-like multiple imputation method.
Time Frame: Baseline to Week 56
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 257 | 254 | 250
kilogram | -2.87 (0.64) | -3.04 (0.67) | -2.81 (0.66)

3. Secondary Outcome: Number of Participants With HbA1c < 7.0 %
Description: Participants who had no available assessment for HbA1c at Week 56 were considered as non-responders.
Time Frame: Week 56
Population: Analysis was performed on mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 257 | 254 | 250
Participants | 155 | 157 | 150

4. Secondary Outcome: Change From Baseline to Week 56 in Fasting Plasma Glucose (FPG)
Description: as for outcome 2
Time Frame: Baseline to Week 56
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 257 | 254 | 250
millimoles per liter (mmol/L) | -1.81 (0.15) | -1.57 (0.15) | -1.71 (0.15)

5. Secondary Outcome: Number of Participants With At Least One Hypoglycemic Events (Documented Symptomatic Hypoglycemia <3.0 mmol/L [<54 mg/dL], Severe Hypoglycemia)
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <54 milligrams per deciliter (mg/dL) (<3.0 mmol/L). Severe hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Baseline up to Week 56
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 313 | 292 | 302
Participants
  Documented symptomatic hypoglycemia (<54 mg/dL) | 3 | 1 | 0
  Severe hypoglycemia | 0 | 0 | 0

6. Secondary Outcome: Number of Hypoglycemic Events (Documented Symptomatic Hypoglycemia <3.0 mmol/L [<54 mg/dL] and Severe Hypoglycemia) Per Participant-Year
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <54 mg/dL (<3.0 mmol/L). Severe hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
Time Frame: Baseline up to Week 56
Population: Analysis was performed on safety population.
Measure: Number; unit: events per participant-year
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
Number analyzed (Participants) | 313 | 292 | 302
events per participant-year
  Documented symptomatic hypoglycemia (<54 mg/dL) | 0.01 | 0.01 | 0
  Severe hypoglycemia | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent up to end of study. Time frame for reporting of treatment emergent adverse events (TEAEs) was from first dose up to 30 days after the last injection of the Investigational Medicinal Product (IMP) (Week 60).
Description: TEAEs were defined as AEs that developed or worsened during the treatment-emergent period. Analysis was performed on safety population.
Arm/Group | Efpeglenatide 4 mg | Efpeglenatide 6 mg | Dulaglutide 1.5 mg
All-Cause Mortality (participants affected / at risk) | 0/313 | 0/292 | 1/302
Serious Adverse Events (participants affected / at risk) | 20/313 | 23/292 | 20/302
Other Adverse Events (participants affected / at risk) | 202/313 | 180/292 | 178/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efpeglenatide 4 mg (N=313) | Efpeglenatide 6 mg (N=292) | Dulaglutide 1.5 mg (N=302)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Spinal Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (3)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Node Dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive Urgency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Omental Necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis Chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Subcapsular Renal Haematoma (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efpeglenatide 4 mg (N=313) | Efpeglenatide 6 mg (N=292) | Dulaglutide 1.5 mg (N=302)
Upper Respiratory Tract Infection (Infections and infestations) | 21 (24) | 18 (20) | 20 (22)
Decreased Appetite (Metabolism and nutrition disorders) | 38 (39) | 50 (56) | 36 (40)
Dizziness (Nervous system disorders) | 18 (18) | 10 (15) | 10 (11)
Abdominal Pain (Gastrointestinal disorders) | 24 (32) | 30 (39) | 16 (25)
Abdominal Pain Upper (Gastrointestinal disorders) | 22 (22) | 16 (20) | 18 (18)
Constipation (Gastrointestinal disorders) | 32 (33) | 34 (37) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 93 (128) | 83 (120) | 90 (134)
Dyspepsia (Gastrointestinal disorders) | 26 (30) | 17 (18) | 15 (20)
Nausea (Gastrointestinal disorders) | 85 (116) | 83 (109) | 78 (111)
Vomiting (Gastrointestinal disorders) | 41 (57) | 45 (65) | 37 (64)
Lipase Increased (Investigations) | 27 (34) | 19 (22) | 24 (29)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor on 09 September 2020. Due to early termination of the study, model-based efficacy analyses were performed in the mITT population instead of the ITT population originally planned and data was carefully considered given that the study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03684642/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT03684642/SAP_001.pdf